CLINICAL TRIAL: NCT00114465
Title: Randomized, Double-Blind, Placebo-Controlled Study of VSL#3 Versus Placebo in the Maintenance of Remission in Crohn's Disease
Brief Title: VSL#3 Versus Placebo in Maintenance of Remission in Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orphan Australia (Other)
Responsible Party: Ian lawrance, Fremantle Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VSL#3Freo
Record Dates: First submitted 2005-06-14; First posted 2005-06-15 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Crohn's Disease
Keywords: Randomized; Double-Blind; Probiotic; Remission; Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VSL#3 (Experimental): Probiotic
  Interventions: Drug: VSL#3
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VSL#3 — VSL#3 1 sachet twice a day
  Arms: VSL#3
Other: Placebo — Placebo 1 sachel twice a day
  Other Names: Blacebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to compare the efficacy of the probiotic VSL#3 versus placebo, in addition to standard maintenance drugs, in maintaining remission in Crohn's disease (CD).

The secondary objectives are:

* To determine the time till flare of CD patients on VSL#3 compared to placebo.
* To assess whether concurrent therapy with VSL#3 leads to an improvement in the quality of life (QOL).
* To assess whether concurrent therapy with VSL#3 reduces the severity of a flare if it occurs.

DETAILED DESCRIPTION:
Advancing knowledge regarding the biology of Crohn's Disease (CD) has identified that the host's innate immunity may impact on the development of intestinal inflammation. Pattern recognition receptors and the Toll-like receptors are able to detect both gram positive and gram negative bacteria, yeasts and flagellin and respond by activation of the innate immune system. By identification of the unmethylated CpG dinucleotide sequences found in bacteria, lymphocytes are stimulated, proinflammatory cytokines like interleukin (IL)-12 and the interferons are induced, and both the mucosal and host defences against the invading pathogens are increased.

A body of evidence from clinical and experimental observations indicates a role for endogenous digestive microflora in the pathogenesis of inflammatory bowel disease (IBD). The distal ileum and the colon are the areas with highest luminal bacterial concentrations and represent the sites of inflammation in IBD. Probiotics have been shown to reduce intestinal inflammation in animal studies. In the human, probiotics may also reduce inflammation particularly in Crohn's disease (CD) and ulcerative colitis (UC). Probiotics are effective in the treatment of acute pouchitis and its prevention. Their use also appears to have some effect in the management of active intestinal inflammation in UC and preliminary results suggest a role in the maintenance of remission.

NOD-2/CARD-15 is a gene that identifies colonic bacteria and can activate the NF-kb pathway in order to destroy the invading bacteria. The identification that mutation of the NOD-2/CARD-15 gene increases a person's susceptibility to developing CD suggests that a defect in the innate immunity may impact on the development of the chronic intestinal inflammation. CD patients are also more likely to have an increase in the mucosal permeability, thus allowing colonic bacteria to cross into the mucosal layer. A central role for the colonic bacteria would thus appear to be possible in the development and maintenance of intestinal inflammation and thus the potential effects and benefits of probiotics in the management of CD requires further investigation.

It appears that treatment with high-potency probiotic preparations for oral bacteriotherapy may enhance the concentrations of protective bacteria of the endogenous digestive microflora and therefore may provide a therapeutic benefit in patients with CD.

This is a phase IV multicentre, randomised, double-blind, placebo-controlled trial of VSL#3 versus placebo in the maintenance of remission in patients with CD. The patients will be randomised to a treatment group receiving one sachet of VSL#3 twice a day, and a group receiving the placebo drug in one sachet twice a day. The patients are assessed at baseline and every 12 weeks until the completion of the study at 52 weeks. At every visit the patient will have routine blood tests for CD, a physical examination and questionnaire will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have a definitive diagnosis of colonic CD or small bowel and colonic CD based on clinical, radiological, endoscopic and pathological findings.
* Subjects should have a CDAI score <150 at week 0
* Patients receiving the following treatment are eligible:

  5 aminosalicylates, if the dose remained constant for 4 weeks before the screening visit and had been used continuously for 8 weeks before screening and the patient has previously flared whilst on the medication; Azathioprine/6MP, if the dose remained constant for 8 weeks prior to the screening visit and had been used continuously for 12 weeks before screening and the patient has previously flared whilst on the medication. Proprietary probiotic preparations must be stopped at least two weeks prior to starting the trial preparation.
* Concomitant use of any other immunosuppressant eg. Methotrexate, tacrolimus, cyclosporine, mycophenolate mofetil, must be at a stable dose of 8 weeks continuous use for 12 weeks prior to screening and the patient has previously flared whilst on the medication.
* Subjects must demonstrate their willingness to participate in the study and comply with the proceedings by signing a written informed consent.
* Men and women ≥18 to < 75 years of age of any race and gender
* Subjects must be free of any clinically significant disease, other than Crohn's disease, that would interfere with the study's evaluations.
* Subjects should understand and be able to adhere to the dosing and visit schedules; and agree to record symptom severity scores, medication times, concomitant medications and adverse events accurately and consistently in a daily diary.

Exclusion Criteria:

Patients should not be enrolled into the study if they meet any of the following criteria:

* Patients with Ulcerative colitis
* Patients with fistulising CD or isolated small bowel CD
* Patients with a CDAI ≥150 at week 0
* Patients on prednisone, budesonide or any form of corticosteroids for the treatment of CD.
* Patients who are incapacitated, largely or wholly bed-ridden or confined to wheelchair, and who have little or no capacity for self-care
* Symptomatic stenosis or ileal strictures.
* Short bowel syndrome
* Serious infections, such as hepatitis, pneumonia, pyelonephritis in the previous 3 months. Less serious infections in the previous 3 months, such as acute upper respiratory tract infection (colds) or uncomplicated urinary tract infection need not be considered exclusions at the discretion of the investigator.
* Documented HIV infection.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, haematological, endocrine, pulmonary, cardiac, neurological or cerebral disease.
* Any currently known malignancy or pre-malignant lesions or any history of malignancy within the past 5 years.
* Patients with alcoholism, alcoholic liver disease, or other chronic liver disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to compare the efficacy of the probiotic VSL#3 versus placebo, in addition to standard maintenance drugs, in maintaining remission in Crohn's disease (CD) | 2 years

SECONDARY OUTCOMES:
Time till flare of CD | within 1 year of commencing therapy
To assess whether concurrent therapy with VSL#3 leads to an improvement in the quality of life | within 1 year of commencing therapy
To assess whether concurrent therapy with VSL#3 reduces the severity of a flare if it occurs | within 1 year of commencing therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ian C Lawrance, MD PhD, Principal Investigator — School of Medicine and Pharmacology, University of Western Australia, Fremantle Hospital
Locations (1):
- Fremantle Hospital, Fremantle, Western Australia, Australia

REFERENCES:
- [Background] Rachmilewitz D, Katakura K, Karmeli F, Hayashi T, Reinus C, Rudensky B, Akira S, Takeda K, Lee J, Takabayashi K, Raz E. Toll-like receptor 9 signaling mediates the anti-inflammatory effects of probiotics in murine experimental colitis. Gastroenterology. 2004 Feb;126(2):520-8. doi: 10.1053/j.gastro.2003.11.019. PMID 14762789
- [Background] Gionchetti P, Rizzello F, Helwig U, Venturi A, Lammers KM, Brigidi P, Vitali B, Poggioli G, Miglioli M, Campieri M. Prophylaxis of pouchitis onset with probiotic therapy: a double-blind, placebo-controlled trial. Gastroenterology. 2003 May;124(5):1202-9. doi: 10.1016/s0016-5085(03)00171-9. PMID 12730861
- [Background] Gionchetti P, Amadini C, Rizzello F, Venturi A, Poggioli G, Campieri M. Diagnosis and treatment of pouchitis. Best Pract Res Clin Gastroenterol. 2003 Feb;17(1):75-87. doi: 10.1053/bega.2002.0348. PMID 12617884
- [Background] Gionchetti P, Amadini C, Rizzello F, Venturi A, Campieri M. Review article: treatment of mild to moderate ulcerative colitis and pouchitis. Aliment Pharmacol Ther. 2002 Jul;16 Suppl 4:13-9. doi: 10.1046/j.1365-2036.16.s4.3.x. PMID 12047254
- [Background] Secondulfo M, de Magistris L, Fiandra R, Caserta L, Belletta M, Tartaglione MT, Riegler G, Biagi F, Corazza GR, Carratu R. Intestinal permeability in Crohn's disease patients and their first degree relatives. Dig Liver Dis. 2001 Nov;33(8):680-5. doi: 10.1016/s1590-8658(01)80045-1. PMID 11785714